CLINICAL TRIAL: NCT04626986
Title: Comparison of Ultrasound Guided Percutaneous Microwave Ablation With Breast Conserving Surgery for Breast Tumor
Brief Title: Comparison of Microwave Ablation With Breast Conserving Surgery for Breast Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Director, Clinical Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2020-09
Record Dates: First submitted 2020-09-27; First posted 2020-11-13 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Breast Tumor; Microwave Ablation; Breast Conserving Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microwave ablation (Experimental): Microwave ablation（MWA）refers to all electromagnetic methods of inducing tumor destruction by using devices with frequencies greater than or equal to 900MHz. The rotation of dipole molecules accounts for most of the heat generated during MWA. Water molecules as dipoles attempt to continuously reorient at the same rate in microwave's oscillating electric field. As a result of microwave transmission, the water molecules flip back and forth billions of times a second. The vigorous movement of water molecules produce friction and heat, thus inducing cellular death via coagulation necrosis. The microwave unit (KY-2000, Kangyou Medical, Nanjing, China) is capable of producing 100 Watts of power at 2450 MHz.The needle antenna has a diameter of 1.6 mm (16G) and a length of 10 cm. The active tip length is 3mm and 5mm.
  Interventions: Procedure: microwave ablation
- breast conserving surgery (Active Comparator): Breast-conserving surgery refers to the removal of the primary tumor and adjacent breast tissue, supplemented by postoperative radiotherapy.Its principle is to remove the primary tumor completely while meet patient's cosmetic satisfaction.The combined treatment of early breast cancer with radiotherapy and chemotherapy is the same as radical surgery or modified radical surgery in terms of local and regional control rate and long-term survival rate. Breast conserving surgery and postoperative comprehensive treatment have become one of the main methods for the treatment of early breast cancer.
  Interventions: Procedure: breast conserving surgery

INTERVENTIONS:
Procedure: microwave ablation — Microwave ablation has the advantages of aesthetics, precise positioning, minimally invasive and painless for patients with early breast cancer.The tumor can be completely killed without injurying adjacent tissue. Some studies have suggested MWA is a safe and effective therapy for the treatment of breast cancer.
  Arms: microwave ablation
Procedure: breast conserving surgery — The treatment of early-stage breast cancer tends to be less-invasive including less morbidity, shorter hospitalization, and improved cosmetic results. Many reports have concluded that there was no difference between breast-conserving surgery and the traditional radical mastectomy for early stage breast cancer in time to distant metastases or overall survival, so breast-conserving surgery is becoming an alternative treatment for early-stage breast cancer.
  Arms: breast conserving surgery

SUMMARY:
The investigators will perform this study to prospectively compare the clinical outcome after percutaneous microwave ablation(MWA) and breast conserving surgery of benign and malignant breast lesion under ultrasound (US) guidance.

DETAILED DESCRIPTION:
A total of more than 300 patients diagnosed with breast tumor in multiple centers will be recruited in this study and underwent US-guided percutaneous MWA and breast conserving surgery treatment. Information for each patient includes demographics; longest diameters of tumors; tumor numbers; tumor pathological type; location of tumor according to whether adjacent to skin, pectoralis, areola and papilla. Ablation variables including session, puncture, time, and power; complete ablation, complications; reduction in volume, palpability, pain and cosmetic satisfying outcomes,recurrence,survival will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. women,
2. with invasive ductal carcinoma of the breast according to core-needle
3. tumor measuring 50mm or smaller, no axillary lymph node metastasis or Ipsilateral grade I and II axillary lymph node metastasis, movable(pT0-2N0-1M0 )
4. located at least 10 mm from the skin surface and chest wall.

Exclusion Criteria:

1. men
2. women who were pregnant or breastfeeding
3. radiologic suspicion of multifocality or extensive intraductal carcinoma
4. histologic diagnosis of lobular carcinoma
5. neoadjuvant therapy
6. previous surgery or radiation therapy of the ipsilateral breast.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
overall survival：Defined as the length of time from the beginning of treatment to death or the last follow-up (if no death) | 5 years
  Defined as the length of time from the beginning of treatment to death or the last follow-up (if no death)
cosmetic satisfaction：Patients are rated whether they are satisfied with the surgical scars（bad / moderate /good / very good） | 3 years
  Patients are rated whether they are satisfied with the surgical scars（bad / moderate /good / very good）

SECONDARY OUTCOMES:
local tumor progress：Defined as the proportion of patients with active tumor at the edge of the treatment ：Defined as the proportion of patients with active tumor at the edge of the treatment | 5 years
  Defined as the proportion of patients with active tumor at the edge of the treatment area during follow-up after the tumor was completely treated
metastasis：Defined as the proportion of cases with metastasis from the beginning of the study to the end of the study or the death of the patient | 5 years
  Defined as the proportion of cases with metastasis from the beginning of the study to the end of the study or the death of the patient
complication：Defined as numbers of participants with side effect and major complications to the end of the study or the death of the patient | 5 years
  Defined as numbers of participants with side effect and major complications to the end of the study or the death of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China